CLINICAL TRIAL: NCT05206058
Title: To Exam the Effects of Phyllanthus Niruri Extracts (Corilagin, Phyllanthin and Brevifolin) on Human Neutrophils
Brief Title: To Exam the Effects of Phyllanthus Niruri Extracts on Human Neutrophils
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202002189B0
Record Dates: First submitted 2022-01-23; First posted 2022-01-25 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2022-01

CONDITIONS: Neutrophil; Phyllanthus Abnormis Poisoning
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Seperation of human neutrophils were according to a standardized procedures and following steps: using 3%(w/v) dextran sedimentation for 30 min, then gradient centrifugation in Ficoll-Hypaque, and hypotonic lysis of erythrocytes. The purified neutrophils were determined by the Trypan blue exclusion method and need to contained >98% viable cells. Then they were suspended in without calcium ion HBSS buffer (pH 7.4), and stored at 4 °C for analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: venipuncture — Plan to enroll 240 health people who are 20-35 years of age. People with received veinpuncture. Blood will be collected at time and drawn into Heparin-coated tube.

SUMMARY:
To exam the effects of Phyllanthus niruri extracts(corilagin, phyllanthin and brevifolin) on human neutrophils

DETAILED DESCRIPTION:
Phyllanthus niruri extracts have anti-inflammatory effects in various cellular systems (monocytes, neutrophil). However, the underlying effects and mechanisms of Phyllanthus niruri extracts on neutrophils have not yet been investigated in detail.

In this study, first we would like to systemic exam the effects of corilagin, phyllanthin and brevifolin, three major active components, on human neutrophils.

Further to clarify whether Phyllanthus niruri extracts have any effect on neutrophils that may provide some insights on the ability of these compounds to modulate the innate immune response in acute organ injury.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers who aged 20-35 years.
* Do not have coagulopathy, systemic infection disease and severe liver and renal function impairment
* Accept venipuncture

Exclusion Criteria:

* Healthy volunteers who aged over 35 years.
* Have coagulopathy, systemic infection disease and severe liver and renal function impairment

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Voluntary healthy donor (20-35 years old) do not have coagulopathy, systemic infective disease and severe liver and renal function impairment.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Measurement of superoxide anion release | After neutrophil isolation, an average of 3 months
  Superoxide anion released from human neutrophils were determined by measuring ferricytochrome c reduction.The neutrophils were activated with fMLF (30 nM) and cytochalasin B(0.5 μg/mL) (fMLF/CB). Changes in absorbance that occurred at 550 nm were observed continuously using a double beam spectrophotometer. Superoxide anion level was calculated using the methods described in previous report.
Measurement of intracellular ROS formation | After neutrophil isolation, an average of 3 months
  Neutrophil ROS production was determined from the conversion of non-fluorescent DHR 123 to fluorescent rhodamine 123, detected using flow cytometry. Neutrophils (2 × 106 cells/ml) were incubated with DHR 123 (2 μM) for 15 min at 37°C, and then treated with honokiol (0.1-10 μM) for 5 min before the addition of fMLP/CB (0.5 μg/ml) for a further 5 min. The change in fluorescence was analysed using flow cytometry

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan